CLINICAL TRIAL: NCT06134713
Title: Effect of Intra-Canal Cryotherapy on Post Operative Pain After Primary and Secondary Root Canal Treatment: A Randomized Controlled Trial
Brief Title: Effect of Intra-Canal Cryotherapy on Postoperative Pain After Endodontic Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajman University (Other)
Collaborators: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Firas Elmsmari, Principal Investigator, Ajman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-F-H-30-NOV
Record Dates: First submitted 2023-11-04; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Endodontically Treated Teeth; Post Operative Pain
Keywords: Root Canal Treatment; Post Operative Pain; Cryotherapy; Nonsurgical Root Canal Retreatment
MeSH Terms: conditions — Tooth, Nonvital; Pain, Postoperative | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Root canal treatment cryotherapy group (Experimental): Conventional root canal treatment with final irrigation using sterile saline at 2.5ºC
  Interventions: Drug: cryotherapy with sterile saline at 2.5ºC
- Root canal RE-treatment cryotherapy group (Experimental): Conventional root canal RE-treatment with final irrigation using sterile saline at 2.5ºC
  Interventions: Drug: cryotherapy with sterile saline at 2.5ºC
- Root canal treatment control group (Active Comparator): Conventional root canal treatment with final irrigation using sterile saline at room temperature
  Interventions: Drug: control with sterile saline at room temperature
- Root canal RE-treatment control group (Active Comparator): Conventional root canal RE-treatment with final irrigation using sterile saline at room temperature
  Interventions: Drug: control with sterile saline at room temperature

INTERVENTIONS:
Drug: cryotherapy with sterile saline at 2.5ºC — In the cryotherapy (experimental group), final irrigation will be performed with 5 ml of 0.9% physiological sterile saline kept refrigerated at 2.5ºC and will be delivered for 1 or 4 minutes with a side vented needle inserted at working length for each canal.
  Arms: Root canal RE-treatment cryotherapy group; Root canal treatment cryotherapy group
Drug: control with sterile saline at room temperature — In the control group, final irrigation will be performed with 5 ml of 0.9% physiological sterile saline kept at room temperature and will be delivered for 1 or 4 minutes with a side vented needle inserted at working length for each canal.
  Arms: Root canal RE-treatment control group; Root canal treatment control group

SUMMARY:
The goal of this randomised clinical trial is to evaluate the effect of cryotherapy on postoperative pain after primary and secondary root canal treatment. The main question[s] it aims to answer are:

* Dose cryotherapy help reduce postoperative pain after primary root canal treatment.
* Dose cryotherapy help reduce postoperative pain after secondary root canal treatment.

Participants will be randomly divided to receive either cryotherapy or irrigation with normal saline and the effect between the two groups in terms of postoperative pain will be compared after primary and secondary root canal treatment.

DETAILED DESCRIPTION:
Procedure

Previous pain assessment:

Both pre- and postoperative pain will be assessed using Huskinsson's visual analog scale (VAS). According to the quantitative data obtained from the VAS scale, these values are categorized as follows: no pain (0), slight pain (0.1-3.9), moderate pain (4-6.9) or pain severe (7-10).

Informed consent After the procedure is carefully explained to the patient and the patient has accepted the treatment plan and signed the Consent, they will be included in the study. Students will give a complete explanation of the study, the forms of pain and how to properly fill out the pain form. If the patient wishes to participate, they will sign the document in order to continue with the treatment and be included in the study.

Root canal treatment and retreatment Vitality test which includes cold test using Endo Ice (Coltene, Switzerland) and Electrical pulp test (EPT) (Shadental, India) for cases of primary root canal treatment. Vertical and lateral percussion tests, periodontal probing, and periapical and bitewing radiographs will be performed in order to perform the pulpal and periapical diagnosis.

The general treatment protocol will be the same for all groups. In case of primary root canal treatment, after the clinical examination, the cold test (Endo-Frost, Coltene-Whaledent, Langenau, Germany) will be used to determine the vitality of the pulp, which will be verified by the presence or absence of bleeding from the root canals during the preparation of the pulp endodontic access.

Local infiltration with 2% lidocaine with epinephrine 1: 80,000 (Ultracain, Normon) will be performed, and absolute isolation with a rubber dam and the department's endodontic protocol will be followed. Access cavity with sterile round diamond drills and Endo-Z drills (Dentsply Maillefer, Ballaigues, Switzerland). The working length (WL) is established with a #10 K-file and apex locator and confirmed with a periapical radiograph. In case of secondary root canal treatment, gutta percha removal and disobturation will be done using different types of rotary and manual files and canals will be negotiated till patency is achieved in all canals, if patency is not achieved the case will be excluded from the study. After which for both primary and secondary root canal treatment instrumentation of the canals will be performed in which they will be irrigated with 1.3% NaOCl solution using a plastic syringe and side-exit needle (Max-i-probe, Kerr-Hawe, Bioggio, Switzerland). Apical patency will be maintained throughout the procedure. Once the procedure is complete, 1 ml of 17% EDTA will be used and a final irrigation with 1.3% NaOCl will be performed with ultrasonic activation using the Irrisafe tip (Acteon, UK).

In the control group, a final irrigation will be performed with 5 ml of 0.9% physiological saline (Sodium Chloride IV infusion 0.9% (Gulf Inject LLC)) at room temperature and in the experimental group with the saline at 2.5ºC for 4 minutes with an endo needle inserted at working length. The saline solution for the control group will be kept at room temperature. The saline solution of the experimental groups will be kept in a refrigerator set at 2.5 C until clinical use.

* Group 1: Conventional root canal treatment with final irrigation with saline at room temperature (n=30).
* Group 2: Conventional root canal retreatment with final irrigation with saline at room temperature (n=30).
* Group 3: Conventional root canal treatment with final irrigation with saline at 2.5ºC for 4 minutes (n=30).
* Group 2: Conventional root canal retreatment with final irrigation with saline at 2.5ºC for 4 minutes (n=30).

The canals will be dried with paper points. The canals of both groups will be filled using a warm gutta-percha filling technique. AH-Plus cement (Dentsply, DeTrey GmbH, Konstanz, Germany) will be used as root canal sealer. Each coronal access will be sealed with a flowable resin (Tetric, IvoclarVivadent AG, SchaanFurstentum, Liechtenstein) and the access cavity will be filled with Glass Ionomer Cement (GIC, ESPE dental, Seefeld, Germany).

Post-operative pain assessment A sheet will be given to the patient with different lines of VAS so that the patient reports the intensity of pain or its absence in the same way that he has been previously taught with preoperative pain at 8, 24 and 48h, 7 days. An ibuprofen 600 mg every 8-12 hours will be recommended for pain control when necessary. The type of analgesic, its quantity and dose will also be recorded in the event that the patients take any type of medication. Patients will be asked to return the VAS collection sheet at the next restoration or general treatment plan continuation visit at the University Clinic. Both the preoperative and postoperative pain results recorded on the Huskinsson VAS scale will be measured by an operator independent of the study, who will be previously calibrated, teaching the evaluator to measure 10 times with a ruler the distance between the initial point of the line to the point marked by the patient on it.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Patients who demonstrate understanding of the study and willingness to participate as evidenced by signing the voluntary informed consent and who received a signed and dated copy of the informed consent form.
* Patients who understand and are willing to comply with all study procedures and restrictions.
* Absence of clinically significant and relevant abnormalities in the clinical history or oral examination.
* Endodontic treatment considered the treatment of choice for both multi and single rooted teeth.
* Endodontic retreatment considered the treatment of choice only in posterior molar teeth (multirooted).
* Only one treatment per patient.

Exclusion Criteria:

* Patients who are allergic to any of the materials used in the treatment.
* Patients with heart pacemaker.
* Patients with any general pathology that requires antibiotic prophylaxis.
* Root resorption, root fractures, impossibility of restoration.
* Pregnant patients.
* Patients who took painkillers in the last 6 hours.
* Case where apical patency couldn't be achieved
* Cases where final obturation quality is compromised.
* Any intra operative factor that complication that can compromise the treatment outcome like root perforation or fractured instrument or inability to localize/prepare any canal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain assessment using the visual analog scale (VAS) | Preoperative, 6 hours,12 hours, 24 hours, 48 hours, 72 hours, 5 days and 7 days
  Both pre- and postoperative pain will be assessed using the visual analog scale (VAS). According to the quantitative data obtained from the VAS scale (from 1 to 10), these values will be categorized as follows: no pain (0), slight pain (0.1-3.9), moderate pain (4-6.9) or severe pain (7-10)

CONTACTS AND LOCATIONS:
Overall Officials: Firas H Elmsmari, PhD, Principal Investigator — Ajman University - College of Dentistry
Locations (1):
- Ajman University, Ajman, United Arab Emirates